CLINICAL TRIAL: NCT07367009
Title: The Effect of the Combination of Adductor Canal Block and Anterior Femoral Cutaneous Nerve Block on Postoperative Inflammatory Biomarkers in Total Knee Arthroplasty
Brief Title: Effect of Combined Adductor Canal and AFCN Block on Postoperative Inflammation
Status: Not yet recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Taşçı, resident doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRH-ST-01
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Anthroplasty
Keywords: total knee arthroplasty; adductor canal block; anterior femoral cutaneous nerve block; postoperative analgesia; inflammatory biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who peripheral nerve block applied: patients who adductor canal block and anterior femoral cutaneous nerve block applied
- patients without peripheral nerve block: patients who do not receive adductor canal block and anterior femoral cutaneous nerve block

SUMMARY:
The aim of this thesis is to evaluate the effects of adding an anterior femoral cutaneous nerve (AFCN) block to the adductor canal block used for postoperative analgesia after total knee arthroplasty on the postoperative inflammatory response, as assessed by inflammatory biomarkers including NLR, PLR, AISI, and CAR.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a common and effective surgical intervention for advanced-stage knee osteoarthritis. However, postoperative pain remains a significant issue affecting the recovery process, opioid requirements, and patient satisfaction. Tissue injury resulting from surgical trauma triggers an inflammatory response that leads to pain. During this process, released mediators activate nerve endings, and the severity of inflammation is generally correlated with pain intensity.

Multimodal analgesia strategies are widely used for postoperative pain management. Peripheral nerve blocks reduce pain scores and opioid consumption, thereby facilitating early mobilization. The adductor canal block is a commonly used technique after knee surgery, providing analgesia to the anteromedial region of the knee while preserving quadriceps muscle strength. However, this block may not adequately anesthetize the anterior femoral cutaneous nerve (AFCN), which innervates the anterior aspect of the thigh. Therefore, an anterior femoral cutaneous nerve block is routinely added to the adductor canal block to improve control of anterior knee pain.

Recent studies have demonstrated that regional anesthesia techniques reduce the inflammatory response, as reflected by biomarkers such as the neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR). This reduction in inflammatory markers has been shown to attenuate the surgical stress response and accelerate wound healing. However, the number of studies evaluating the effects of peripheral nerve blocks on biomarkers such as NLR, PLR, aggregate index of systemic inflammation (AISI), and C-reactive protein/albumin ratio (CAR) in knee surgery remains limited.

In our clinic, the choice of anesthesia technique in daily practice is determined based on the surgical site, type of procedure, patient positioning, and the experience of the anesthesia team. In patients undergoing total knee arthroplasty, ultrasound-guided adductor canal block combined with an anterior femoral cutaneous nerve block is routinely performed for postoperative pain management. The efficacy and safety of both blocks have been demonstrated in regional anesthesia guidelines and previous studies.

The primary outcome of this observational study is to evaluate the effect of adding an anterior femoral cutaneous nerve block to the adductor canal block on the inflammatory response, as assessed by biomarkers such as NLR, PLR, AISI, and CAR, in patients undergoing total knee arthroplasty. Secondary outcomes include postoperative opioid consumption, incidence of nausea and vomiting, early mobilization, and wound healing.

In our clinic, both general and regional anesthesia techniques are applied for knee arthroplasty according to patient suitability. Among regional anesthesia techniques, spinal anesthesia and peripheral nerve blocks are routinely preferred for both anesthesia and analgesia management based on the decision of an experienced anesthesiologist.

This study was designed as a prospective observational study and will be conducted at Fatih Sultan Mehmet Training and Research Hospital between January 2026 and January 2027 following approval by the local ethics committee. Patients aged 18 years or older, scheduled for elective unilateral total knee arthroplasty under spinal anesthesia (SA), classified as American Society of Anesthesiologists (ASA) physical status I-III, and who provide written informed consent after being informed one day before surgery on the ward will be included. Based on a power analysis performed using G*Power version 3.1.9.4 with a power of 80% and a type I error rate of 5%, a total of 60 patients is planned to be enrolled.

Exclusion criteria include emergency surgery; revision or bilateral procedures; general anesthesia or conversion to general anesthesia due to failed regional block; body mass index (BMI) ≥35 kg/m²; ASA physical status >III; local infection, hematoma, previous surgery, or deformity at the block site; coagulation disorders; history of hematologic, renal, or hepatic disease; advanced respiratory or cardiac failure; malignancy; anticoagulant therapy; history of local anesthetic allergy or toxicity; impaired cooperation; Alzheimer's disease; dementia; psychiatric or neurological disorders; language or communication barriers; chronic analgesic use; chronic alcohol consumption; substance abuse; and refusal to participate.

Demographic data (age, sex, ASA status, BMI), comorbidities, and routinely assessed preoperative laboratory parameters-including hemoglobin, hematocrit, white blood cell count (WBC), platelet count, PLR, NLR, C-reactive protein (CRP), and albumin levels-will be recorded for all included patients. Additionally, the CRP/albumin ratio (CAR) and the aggregate index of systemic inflammation (AISI = platelet × neutrophil × monocyte / lymphocyte) will be calculated and documented.

Upon arrival in the operating room, standard monitoring-including electrocardiography (ECG), noninvasive blood pressure, peripheral oxygen saturation (SpO₂), and body temperature-will be applied. Following monitoring and premedication with intravenous midazolam (0.02 mg/kg), spinal anesthesia will be performed. Under sterile conditions in the sitting position, a 25-gauge spinal needle will be inserted at the L3-L4 interspace. After confirmation of clear cerebrospinal fluid flow, 15 mg of 0.5% hyperbaric bupivacaine will be injected. Patients will then be placed in the supine position, and sensory block level (pinprick test) and motor block (Bromage score) will be assessed. Surgery will be initiated in patients achieving a sensory block at or above the T12 level and a Bromage score of 2. Hemodynamic parameters (heart rate, systolic, diastolic, and mean arterial pressure), body temperature, and SpO₂ values will be recorded at 20-minute intervals intraoperatively.

In our clinic, there is no standardized anesthesia or postoperative analgesia protocol; the choice is based on the surgical site, type of surgery, and clinician experience. Following total knee arthroplasty, ultrasound-guided peripheral nerve blocks may be used for postoperative analgesia according to anesthesiologist preference. The combination of adductor canal block and anterior femoral cutaneous nerve block is commonly preferred. At the end of surgery, while the patient is in the supine position, ultrasound-guided adductor canal and AFCN blocks will be performed. For the adductor canal block, 15 mL of 0.25% bupivacaine will be injected around the femoral artery beneath the sartorius muscle at the mid-thigh level. Subsequently, the AFCN block will be completed by injecting 10 mL of 0.25% bupivacaine superficial to the sartorius muscle at the same level. This combination provides effective analgesia for the anterior and medial aspects of the knee while preserving quadriceps muscle strength and allowing early mobilization.

All patients will receive 1 g of intravenous paracetamol as part of standard postoperative analgesia prophylaxis 20 minutes before the end of surgery. At the end of surgery, patient-controlled analgesia (PCA) with tramadol will be prepared using a 15 mg bolus dose and a 20-minute lockout interval and initiated in the post-anesthesia care unit (PACU). Surgery duration, anesthesia duration, and tourniquet time will be recorded.

Postoperatively, patients will be monitored in the PACU. Sensory block level, hemodynamic parameters, SpO₂ values, and pain scores at rest and during movement will be recorded at 0, 15, and 30 minutes in the PACU, and at 2, 4, 8, 12, and 24 hours on the ward. Nausea and vomiting, sedation level, and quadriceps muscle strength will also be documented. Pain intensity will be assessed using the 10-point Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain). Nausea and vomiting severity will be evaluated using a 5-point scale. Patients with an Aldrete score ≥9 and postoperative NRS <4 will be transferred to the ward.

Quadriceps muscle strength will be evaluated as follows: normal strength (score 0), mild weakness (score 1), and severe weakness (score 2). Scores of 1 and 2 will be considered quadriceps weakness.

Postoperative analgesia with tramadol PCA will be continued on the ward. Patients with an NRS score ≥4 will receive 50 mg intravenous dexketoprofen as rescue analgesia. Nausea and vomiting will be treated with intravenous ondansetron and dexamethasone as needed.

Total tramadol consumption, number of PCA demands, time to first rescue analgesic requirement, additional antiemetic use, and block-related complications will be recorded. Laboratory parameters will be recorded at postoperative 12 and 24 hours. Patients will be divided into two subgroups based on receipt of peripheral nerve blocks. Surgical site infection will be evaluated on postoperative days 15 and 30.

This study will document procedures routinely performed in clinical practice and will not impose any additional cost on patients or the institution.

ELIGIBILITY:
Inclusion Criteria:

* • Patients scheduled for elective unilateral total knee arthroplasty under spinal anesthesia

  * Aged 18 years and older
  * Body mass index (BMI) <40 kg/m²
  * ASA physical status I-III
  * Provision of written informed consent

Exclusion Criteria:• Emergency surgery

* Revision or bilateral surgery
* General anesthesia or conversion to general anesthesia due to failed block
* BMI ≥40 kg/m²
* ASA physical status >III
* Local infection, hematoma, previous surgery, or deformity at the block site
* Coagulopathy or history of hematologic, renal, or hepatic disease; advanced respiratory or cardiac failure; malignancy
* Use of anticoagulant therapy
* History of local anesthetic allergy or toxicity
* Impaired cooperation, Alzheimer's disease, dementia, psychiatric or neurological disorders, or language/communication barriers
* Chronic analgesic use, chronic alcohol consumption, or substance abuse
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older, scheduled for elective unilateral total knee arthroplasty under spinal anesthesia (SA), classified as American Society of Anesthesiologists (ASA) physical status I-III, and who provided written informed consent after being informed one day before surgery on the ward, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
assessment of post operative inflammatuar markes | it will be recorded at 0, 15, and 30 minutes in the PACU, and at 2, 4, 8, 12, and 24 hours on the ward.
  The primary objective of this observational study is to evaluate the effect of adding an anterior femoral cutaneous nerve block to the adductor canal block on the inflammatory response, as assessed by biomarkers such as NLR, PLR, AISI, and CAR, in patients undergoing total knee arthroplasty.

SECONDARY OUTCOMES:
postoperative opioid consumption, wound healing | it will be recorded at 0, 15, and 30 minutes in the PACU, and at 2, 4, 8, 12, and 24 hours on the ward.
  The secondary outcomes are to investigate the effects of this block combination on postoperative opioid consumption, the incidence of nausea and vomiting, early mobilization, and wound healing

CONTACTS AND LOCATIONS:
Overall Officials: oznur demiroluk, as prof, Study Director — fatih sultan mehmet traing and research hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Razzaz M.; Youssif G.; Wahba S.; Mohamed S.; Mohamed A. Analgesic efficacy of ultrasound guided anterior femoral cutaneous nerve block (AFCNB) plus femoral triangle block (FTB) vs. adductor canal block (ACB) in total knee arthroplasty, Anaesthesia, Pain & Intensive Care, 2025
- [Result] Domagalska M, Ciftsi B, Janusz P, Reysner T, Kolasinski J, Wieczorowska-Tobis K, Kowalski G. The neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR) levels following erector spinae plane block (ESPB) in posterior lumbar decompression: a randomized, controlled trial. Eur Spine J. 2023 Dec;32(12):4192-4199. doi: 10.1007/s00586-023-07913-z. Epub 2023 Sep 5. PMID 37668689
- [Result] Domagalska M, Reysner T, Kowalski G, Daroszewski P, Mularski A, Wieczorowska-Tobis K. Pain Management, Functional Recovery, and Stress Response Expressed by NLR and PLR after the iPACK Block Combined with Adductor Canal Block for Total Knee Arthroplasty-A Prospective, Randomised, Double-Blinded Clinical Trial. J Clin Med. 2023 Nov 14;12(22):7088. doi: 10.3390/jcm12227088. PMID 38002702